CLINICAL TRIAL: NCT04002037
Title: Differential Efficacy of Corticosteroid Solutions for Non-Operative Treatment of Digit Flexor Tenosynovitis: A Double-Blind Prospective Randomized Clinical Trial
Brief Title: Differential Efficacy of Corticosteroid Solutions for Non-Operative Treatment of Digit Flexor Tenosynovitis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Preliminary analysis revealed no difference
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Daniel London, Assistant Professor, Orthopaedic Surgery, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014039
Record Dates: First submitted 2019-06-21; First posted 2019-06-28 (Actual); Results first posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Trigger Finger
Keywords: Trigger Finger
MeSH Terms: conditions — Trigger Finger Disorder | interventions — Triamcinolone Acetonide; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Triamcinolone 40mg/mL (Active Comparator): A corticosteroid injection of Triamcinolone 40mg/mL will be given to subjects to treat their symptoms of trigger finger.
  Interventions: Drug: Triamcinolone Acetonide 40mg/mL
- Triamcinolone 10mg/mL (Active Comparator): A corticosteroid injection of Triamcinolone 10mg/mL will be given to subjects to treat their symptoms of trigger finger.
  Interventions: Drug: Triamcinolone Acetonide 10mg/mL
- Soluble dexamethasone 4mg/mL (Active Comparator): A corticosteroid injection of Soluble Dexamethasone 4mg/mL will be given to subjects to treat their symptoms of trigger finger.
  Interventions: Drug: Dexamethasone 4 mg/ml

INTERVENTIONS:
Drug: Triamcinolone Acetonide 40mg/mL — Corticosteroid injection will occur up to two times if trigger finger symptoms are not resolved.
  Arms: Triamcinolone 40mg/mL
Drug: Triamcinolone Acetonide 10mg/mL — Corticosteroid injection will occur up to two times if trigger finger symptoms are not resolved.
  Arms: Triamcinolone 10mg/mL
Drug: Dexamethasone 4 mg/ml — Corticosteroid injection will occur up to two times if trigger finger symptoms are not resolved.
  Arms: Soluble dexamethasone 4mg/mL

SUMMARY:
Trigger finger is a common cause of hand pain and dysfunction. Its due to chronic inflammation of the flexor tendon that leads to a pulley system mismatch. Historically it has been managed either conservatively with corticosteroid injections or through a surgical release of the A1 pulley. Several corticosteroids have been used for injection- dexamethasone, methylprednisolone, triamcinolone, betamethasone, paramethasone, etc. The purpose of out study is to determine if a 0.5 cc injection of Triamcinolone 40 mg/mL will be the most effective steroid injection for the non-surgical treatment. Approximately 200 subjects will be enrolled and randomized to one of three treatment arms: Triamcinolone 40mg/mL, Triamcinolone 10mg/mL and Soluble dexamethasone 4mg/mL. Treatment success will be defined as lack of conversion to surgical treatment, or no desire to proceed with surgery during study period (3 months).

DETAILED DESCRIPTION:
Idiopathic stenosing tenosynovitis of the digits, more commonly known as "trigger finger", is a common cause of hand pain and dysfunction. Many previous studies have described the pathophysiology of this condition and it can be summarized as inflammation of the flexor tendons leading to a size mismatch between the tendon and the flexor pulley system. By far the most common location of this mismatch is at the A1 pulley.

The current mainstay of treatment has been:

1. Injection of corticosteroid into the area immediately surrounding the A1 pulley and flexor tendon
2. Surgical release of the A1 pulley

Several corticosteroids have been used for injection- dexamethasone, methylprednisolone, triamcinolone, betamethasone, paramethasone, etc. Less commonly used treatment strategies have included: topical NSAIDs and extracorporeal shock therapy. The typical progression of treatment is one or two steroid injections and then surgical release if injections have failed.

To our knowledge, there have been no head to head comparison studies of the efficacy of different corticosteroid formulations in preventing conversion to surgical treatment. In our study, the investigators will look at the efficacy of two of the most commonly used steroids: triamcinolone and dexamethasone.

Objectives:

Primary outcome: Treatment success, defined as lack of conversion to surgical treatment, or no desire to proceed with surgery during study period (3 months).

Secondary outcomes: Grade of triggering (Green classification of trigger finger severity1), QuickDASH (Disabilities of the Arm, Shoulder and Hand) and PROMIS Upper Extremity scores, VAS.

Inclusion/Exclusion:

Inclusion criteria:

1. Adults aged 18 years and older
2. At least one symptomatic trigger finger
3. Patients recommended to receive corticosteroid injections

Exclusion criteria:

1. Previous surgeries/injections for trigger fingers in digit being treated for study
2. Participating in another clinical trial
3. Inability to receive corticosteroid injections (i.e. allergies, adverse reactions, etc.)
4. Unable to sign informed consent
5. Pregnant or plan to become pregnant

Study Procedures/Methods:

Enrollment/Randomization/Treatment Visit:

Eligible patients presenting with primary flexor tenosynovitis will be enrolled on a voluntary basis. Prior to the injection, subjects will be asked to complete the PROMIS and QuickDASH surveys to collect data at baseline.

Enrolled patients will be randomized to one of three treatment arms:

1. Triamcinolone 40mg/mL
2. Triamcinolone 10mg/mL
3. Soluble dexamethasone 4mg/mL

Each study patient will receive the appropriate corticosteroid injection in the affected digit(s), consisting of a 1:1 mixture of 1% lidocaine plain and corticosteroid, total volume 1cc.

Blinding:

Syringes will be prepared and masked with opaque tape by the clinic nurses, thus providing blinding for providers administering the injection.

Follow-Up/Clinic Visits:

Subjects will be re-evaluated at 6 weeks post-injection and, if still symptomatic, will undergo a second injection of the same corticosteroid solution. At final follow-up (12 weeks), symptomatic patients who have failed treatment after 2 injections will be offered surgical release of the A1 pulley. Subjects who refuse a second injection at 6 weeks follow-up will be offered surgery, and the reason for refusal (treatment failure) will be recorded.

The visits and all research activity will be outlined below:

6 Week Follow-Up:

Objective Measures:

- Grade of triggering (Green classification of trigger finger severity1)

Subjective Measures:

* QuickDASH
* PROMIS scores
* VAS Second Corticosteroid injection (if subject still symptomatic)

  12 Week (3 Month) Follow-Up (if applicable):

Objective Measures:

- Grade of triggering (Green classification of trigger finger severity1)

Subjective Measures:

- QuickDASH

- PROMIS scores

- VAS

6 Month Follow-Up: The patient will be contacted to check on the status of their condition. If they are still experiencing a degree of triggering they will be advised by their physician to return to clinic for a standard of care visit. If they are no longer experiencing triggering, they will be asked to complete a survey over the phone or online only.

Specimen Collection: If a patient is recommended to undergo surgery at the end of the study, the tenosynovium that is normally resected and discarded after surgery will be collected for analysis. After collection these tissues and data will be identified from the patient and assigned a number for use in study analysis. The investigators seek to only collect tissues from patients that are normally removed and discarded during trigger finger release procedures. None of the patients will undergo additional surgical procedures for the collection of tissues in this study. For simplification purposes, potential subjects must agree to the collection of these specimens to participate in the study, even if they do not end up needing surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years and older
2. At least one symptomatic trigger finger
3. Patients recommended to receive corticosteroid injections

Exclusion Criteria:

1. Previous surgeries/injections for trigger fingers in digit being treated for study
2. Participating in another clinical trial
3. Inability to receive corticosteroid injections (i.e. allergies, adverse reactions, etc.)
4. Unable to sign informed consent
5. Pregnant or plan to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2023-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel London, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri Health Care, Columbia, Missouri, United States

REFERENCES:
- [Background] 1- Wolfe SW, Hotchkiss RN, Pederson WC, Kozin SH, Tendinopathy, in: Green's Operative Hand Surgery, 6th edition, Churchill Livingstone, Chap. 62, p. 5, 2011.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Triamcinolone 40mg/mL | Triamcinolone 10mg/mL | Soluble Dexamethasone 4mg/mL
Started | 24 | 43 | 28
Completed | 24 | 43 | 28
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Triamcinolone 40mg/mL | Triamcinolone 10mg/mL | Soluble Dexamethasone 4mg/mL | Total
Number analyzed (Participants) | 24 | 43 | 28 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.54 (9.99) | 63.77 (10.65) | 61.75 (9.11) | 63.37 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 30 | 22 | 69
  Male | 7 | 13 | 6 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 2
  White | 22 | 40 | 28 | 90
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Disabilities of the Arm, Shoulder and Hand (DASH)
Description: The patient will be asked to complete a questionnaire with questions related to their hand. Their answers will be scored on a scale of 0-100 with 0 being no disability and 100 being the highest level of disability.
Time Frame: 6 Weeks
Population: The analysis population differs from the participant flow module due to participants not completing the outcome measure or due to early study termination.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Triamcinolone 40mg/mL | Triamcinolone 10mg/mL | Soluble Dexamethasone 4mg/mL
Number analyzed (Participants) | 12 | 27 | 16
score on a scale | 12.69 (19.87) | 18.69 (18.73) | 24.72 (13.74)

2. Primary Outcome: Disabilities of the Arm, Shoulder and Hand (DASH)
Description: as for outcome 1
Time Frame: 12 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Triamcinolone 40mg/mL | Triamcinolone 10mg/mL | Soluble Dexamethasone 4mg/mL
Number analyzed (Participants) | 13 | 24 | 12
score on a scale | 17.66 (19.88) | 18.09 (17.71) | 23.38 (22.91)

3. Primary Outcome: Disabilities of the Arm, Shoulder and Hand (DASH)
Description: as for outcome 1
Time Frame: 6 Month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Triamcinolone 40mg/mL | Triamcinolone 10mg/mL | Soluble Dexamethasone 4mg/mL
Number analyzed (Participants) | 13 | 30 | 14
score on a scale | 22.73 (19.53) | 22.12 (20.55) | 13.64 (16.24)

4. Primary Outcome: Pain Visual Analog Score (VAS)
Description: The patient will be asked to report their pain on a scale of 0 - 10 using the Visual Analog Scale with 0 being no pain and 10 being the worst pain the patient can imagine.
Time Frame: 6 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Triamcinolone 40mg/mL | Triamcinolone 10mg/mL | Soluble Dexamethasone 4mg/mL
Number analyzed (Participants) | 12 | 27 | 14
score on a scale | 1.08 (2.15) | 1.33 (2.2) | 2.04 (2.09)

5. Primary Outcome: Pain Visual Analog Score (VAS)
Description: as for outcome 4
Time Frame: 12 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Triamcinolone 40mg/mL | Triamcinolone 10mg/mL | Soluble Dexamethasone 4mg/mL
Number analyzed (Participants) | 13 | 24 | 15
score on a scale | 1.15 (1.91) | 2.38 (2.37) | 3.33 (3.22)

6. Primary Outcome: Pain Visual Analog Score (VAS)
Description: as for outcome 4
Time Frame: 6 Month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Triamcinolone 40mg/mL | Triamcinolone 10mg/mL | Soluble Dexamethasone 4mg/mL
Number analyzed (Participants) | 15 | 29 | 16
score on a scale | 1.53 (1.46) | 1.97 (2.41) | 1.38 (2.13)

7. Primary Outcome: Patient Reported Outcomes Measurement Information System (PROMIS) Upper Extremity Scores
Description: PROMIS Physical Function - Upper Extremity is a self-reported performance measure assessing physical function of the upper extremity focusing on nine activities that require use of the upper extremity including shoulder, arm, and hand activities. Responses are as follows: 5 = Without any difficulty; 4 = With a little difficulty; 3=With some difficulty; 2=With much difficulty; and 1=Unable to do.
  The PROMIS Upper Extremity assessment evaluates upper extremity function, with raw scores typically ranging from 8 to 40, depending on the specific form used. These raw scores are converted to T-scores using a standardized table, with a mean of 50 and a standard deviation of 10. These T-scores range from 15 to 61. A higher T-score indicates better upper extremity function, while a lower T-score signifies greater impairment.
Time Frame: 6 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Triamcinolone 40mg/mL | Triamcinolone 10mg/mL | Soluble Dexamethasone 4mg/mL
Number analyzed (Participants) | 12 | 26 | 9
score on a scale | 48.24 (13.45) | 44.49 (11.89) | 37.55 (8.98)

8. Primary Outcome: Patient Reported Outcomes Measurement Information System (PROMIS) Upper Extremity Scores
Description: as for outcome 7
Time Frame: 12 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Triamcinolone 40mg/mL | Triamcinolone 10mg/mL | Soluble Dexamethasone 4mg/mL
Number analyzed (Participants) | 11 | 22 | 14
score on a scale | 48.28 (12.09) | 44.82 (11.68) | 43.44 (12.4)

9. Primary Outcome: Patient Reported Outcomes Measurement Information System (PROMIS) Upper Extremity Scores
Description: as for outcome 7
Time Frame: 6 Month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Triamcinolone 40mg/mL | Triamcinolone 10mg/mL | Soluble Dexamethasone 4mg/mL
Number analyzed (Participants) | 15 | 29 | 14
score on a scale | 38.46 (12.9) | 42.23 (11.43) | 47.9 (11.51)

ADVERSE EVENTS:
Time Frame: Participant follow-up post enrollment was for 6 months.
Description: There is no difference in the definition of adverse event and/or serious adverse event.
Arm/Group | Triamcinolone 40mg/mL | Triamcinolone 10mg/mL | Soluble Dexamethasone 4mg/mL
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/43 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/43 | 0/28
Other Adverse Events (participants affected / at risk) | 0/24 | 0/43 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-27): https://cdn.clinicaltrials.gov/large-docs/37/NCT04002037/Prot_SAP_000.pdf